CLINICAL TRIAL: NCT05794828
Title: Erector Spinae Regional Anesthesia for Pain Control in the Emergency Department
Brief Title: Erector Spinae Regional Anesthesia for Pain Control
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20220911H
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Pain Management
Keywords: Erector spinae plane block; ESPB; Pain reduction
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Single group open label assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Erector Spinae Plane Block (ESP) administration (Experimental): Patients with the listed diagnoses will be offered and then consented for an ESPB under ultrasound guidance.
  Interventions: Drug: Bupivacaine Injection

INTERVENTIONS:
Drug: Bupivacaine Injection — Bucivacaine will be administered intramuscularly according to package insert directions after first numbing the area with lidocaine subcutaneously
  Other Names: Bupivacaine Hydrochloride Injection

SUMMARY:
Interventional study to use erector spinae plane block (ESPB) on diagnoses of posterior or lateral rib fractures, vertebral fractures, pancreatitis, pancreatic cancer, renal colic, and back pain for multimodal pain therapy to determine its assistance with pain relief as well as the patient's use of opiates after block completion

DETAILED DESCRIPTION:
Patients with the listed diagnoses will be offered and then consented for an ESPB under ultrasound guidance. They will rate their pain before and 30 minutes after the procedure using the ordinal categorical data on a numeric pain scale. Total patient opiate use will be gathered up to 8 hours after block completion.

ELIGIBILITY:
Inclusion Criteria:

* Posterior/lateral rib or vertebral fractures
* Pancreatitis or pancreatic cancer
* Renal colic
* Back pain

Exclusion Criteria:

* Unstable vitals
* Infection or open wound over insertion site
* Prior allergic reaction to local anesthetic
* Pregnant females
* Patients <18 years old
* Altered mentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Pain Scale Rating | Baseline to study procedure end (approximately 30 minutes)
  Change in pain scale rating assessed by the participants on a scale from 0-10 with 0 indicating no pain and 10 indicating the most severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Ritz, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (4):
- United States (4):
  - Crozer Chester Medical Center, Ridley Park, Pennsylvania
  - Crozer Chester Medical Center, Upland, Pennsylvania
  - University Hospital, San Antonio, Texas
  - Baylor Scott & White, Temple, Texas

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared in a peer reviewed publication after acceptance by the journal
Supporting Information: Study Protocol, SAP
Time Frame: At study completion, after acceptance into a peer reviewed journal